CLINICAL TRIAL: NCT00311714
Title: CS-8958 - A Phase I, Double-Blind, Placebo-Controlled, Ascending Single Inhaled Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of Biota-CS-8958
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0077; 1833-094
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza, United Kingdom
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Drug: CS-8958 formulated as dry powder
Other: Placebo

SUMMARY:
This study will look at the safety, tolerability and what the body does to CS-8958 given to 40 healthy volunteers 18-55 years old. CS-8958 is a dry-powder investigational drug that is breathed into the lungs through an inhaler device. The researchers will collect information about any problems that volunteers have while taking the drug and about changes in blood pressure and how the heart is working. Volunteers will have breathing tests, physical examinations, and blood samples collected for laboratory tests. The researchers will also look at how much of the medication travels throughout the body versus how much stays only in the lungs. Doses of the medication will be tested at one level and then at higher and higher levels after a safety committee reviews the safety and tolerability information on volunteers prior to the next higher dose being given. Each volunteer will participate for up to 6 weeks from initial screening to the follow up visit and spend 7 days in the clinic.

DETAILED DESCRIPTION:
This study is a phase I, double-blind, placebo-controlled, ascending single inhaled dose, safety, tolerability and pharmacokinetic study of CS-8958 in healthy subjects. CS-8958 is an investigational drug substance, which is formulated as a dry-powder. Capsules of the dry powder are inserted into a FlowCaps® inhaler device. FlowCaps® is a re-fillable, dry-powder, breath-actuated inhaler device, which holds up to 14 capsules. Upon actuation the powder contained in one capsule is delivered to the respiratory tract. The primary study objective is to evaluate the safety and tolerability of CS-8958 (5, 10, 20, and 40 mg) in healthy subjects after a single dose administered via inhalation. Parameters are adverse events (AEs), vital signs including blood pressure/pulse rate (BP/PR) measurements, functional oxygen saturation of arterial haemoglobin (SpO2), electrocardiogram (ECG) examinations, spirometry (Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1), FEV percentage in 1 second (FEV 1%), FEV1/FVC ratio, Forced Expiratory Flow Rate (FEF) 25%-75%, Peak Expiratory Flow Rate (PEFR), physical examinations, mood assessments, and laboratory parameters. The secondary study objective is to assess the systemic exposure of CS-8958 and its active metabolite R-125489 after single inhaled doses of CS-8958 in healthy subjects. At Covance Clinical Research Unit Ltd, Leeds, UK, 40 subjects will be studied in 4 groups (Groups A to D) with each group consisting of 10 subjects. Healthy male and female subjects aged 18-55 years inclusive will be recruited for the study. There will be four investigational product treatment groups (Groups A, B, C, and D). Within each group, subjects will be randomly allocated to Arm 1 or Arm 2. The study product doses will be administered in an escalating manner. The Safety Monitoring Committee (SMC) will review the safety and tolerability data from each group, prior to administration of the next dose. Following these reviews, the dose increment for subsequent groups may be increased, or the doses administered may be reduced, and may be lower than the starting dose. The maximum dose level to be studied will be 40 mg. The primary outcome measures include safety and tolerability. These outcome measures will be addressed in terms of occurrences of treatment-emergent AEs, changes in vital signs including BP and PR, SpO2, oral body temperature, ECG, spirometry (FVC, FEV1, FEV 1%, FEV1/FVC ratio, FEF 25-75% and PEFR), physical examinations, mood assessments, and laboratory parameters. Secondary outcome measures will include pharmacokinetic parameters. These parameters will be calculated for CS-8958 and R-125489 concentrations in plasma and urine using a non-compartmental approach.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 55 years of age. Male subjects should use appropriate contraception (e.g. condoms) during the time interval between dosing until 3 months after dosing. Female subjects should be of non-child bearing potential. Female subjects 50 years of age or less must be surgically sterile or post-menopausal (defined as at least two years post cessation of menses and/or follicle-stimulating hormone (FSH) >18 mIU/mL and serum oestradiol <110 pmol/L), non-lactating and have a negative serum pregnancy test. Female subjects of more than 51 years of age must be surgically sterile or post menopausal (defined by a value of FSH >18 mIU/mL and no spontaneous menstruation for at least one year before investigational product administration), non-lactating and have a negative serum pregnancy test.
* Vital signs within normal limits: systolic BP between 90 and 150 mmHg, diastolic BP between 40 and 90 mmHg, pulse rate between 35 and 100 bpm (confirmed as sinus rhythm if between 35 and 40 bpm), oral temperature between 35.5°C and 37.7°C and oxygen saturation of at least 98%.
* Normal physical examination and laboratory findings. Grade 1 laboratory abnormalities for non-essential tests and clinical findings considered not clinically significant or a variant of normal may be acceptable following discussion between the Investigator and the Sponsor.
* No abnormality in the ECG; specifically QTc <450 ms and PR 120-200 ms.
* None of the following abnormal laboratory findings:
* AST >51 IU/L (males) or >46 IU/L (females) [based on 1.25 x ULN]
* ALT >61 IU/L (males) or >48 IU/L (females) [based on 1.25 x ULN]
* Serum creatinine >104 micro mol/L (males) or >84 micro mol/L (females)
* Glucose <3.8 or >5.5 mmol/L
* Potassium <3.9 or >5.3 mmol/L (males) or <3.8 or >5.4 mmol/L (females)
* Haemoglobin <13.5 or >18.0 g/dL (males) or <11.5 or >16 g/dL (females)
* Platelets <152 or >338 x 10^9/L (males) or <150 or >400 x 10^9/L (females)
* WBC <3.6 or >10.0 x 10^9/L (males) or <4.0 or >11.0 x 10^9/L (females)
* Neutrophils <1.80 x 10^9/L (males) or <2.00 x 10^9/L (females)
* No disease that the Investigator regards as clinically relevant.
* Negative results in Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface antigen (HBsAg) and Hepatitis C antibody tests.
* Individuals who have been registered with a general practitioner within the United Kingdom for at least 3 months before enrollment and whose general practitioners have replied to a medical history questionnaire.
* Individuals who have freely given Informed Consent in writing.
* Able to perform respiratory testing.

Exclusion Criteria:

* Subjects who have taken any prescription medication (with the exception of hormone replacement therapy (HRT)) within 14 days or any non-prescription (with the exception of vitamin/mineral supplements) within the last 7 days prior to the administration of the investigational product (Day 1).
* Intake of any investigational drug within 4 months (new chemical entity) or 3 months (marketed compounds) prior to the intake of investigational product (Day 1).
* History of allergy or serious adverse reaction to the excipient or neuraminidase inhibitor.
* A history or clinical evidence of significant cerebrovascular, cardiovascular, gastrointestinal, or haematological disease, or myocardial infarction, or a previous history of any other serious underlying disease (including immunocompromised subjects and/or neutropenic subjects) that, in the opinion of the Investigator would interfere with the conduct of the study.
* A history or clinical evidence of significant respiratory disease (including asthma, hyper-reactive lung disease, COPD, cystic fibrosis and/or recurrent lower respiratory tract infection) and/or upper respiratory tract infection within the last month or lower respiratory tract infection within the last three months.
* A history or clinical evidence of renal disease (including renovascular occlusive disease), nephrectomy and/or renal transplant, and/or previous clinically significant laboratory abnormalities of renal function parameters. All subjects with serum creatinine outside the normal laboratory reference range at screening and before randomization that are regarded by the Investigator as clinically significant.
* A history or clinical evidence of hepatic disease and/or previous clinically significant laboratory abnormalities of liver function parameters. All subjects with alanine transaminase (ALT) and/or aspartate transaminase (AST) outside the normal laboratory reference range at screening and before randomization, that are regarded by the Investigator as clinically significant. Subjects known to have experienced elevated liver enzyme values in previous clinical studies will also be excluded.
* Psychiatric or emotional problems that would limit the ability of the subject to comply with study requirements.
* Body Mass Index (BMI) <18.5 kg/m squared or >30.0 kg/m squared.
* FEV1 less than or equal to 85%, FEV (1.0%) less than or equal to 70%, and/or FVC less than or equal to 80% of the predicted value, as calculated from standard age and height formula.
* History of alcohol and/or drug abuse (verified by drug screening).
* Receipt of blood or blood products or loss of 450 mL or more of blood during the last three months before screening.
* Unwillingness or inability to provide Informed Consent or to participate satisfactorily for the entire study period.
* Subjects who smoke or have been non-smokers for less than 3 months prior to Screening.
* Subjects who were previously enrolled in this study.
* Subjects who in the opinion of the investigating physician are unable to use the inhaler device after training.
* Poor veins, or fear of venipuncture or sight of blood.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2007-04; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd (Covance CRU), Leeds, United Kingdom